CLINICAL TRIAL: NCT02525029
Title: Phase I/II Study of Human Chorionic Gonadotropin and Epidermal Growth Factor Supplementation (Pregnyl®) to Support Tolerance and Repair As Adjunct Therapy in High-Risk or Refractory Acute Graft-Versus-Host Disease
Brief Title: Study of Pregnyl as Adjunct Therapy for High-Risk or Refractory Acute GVHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014LS020; NCI-2015-02022 (Registry Identifier: CTRP)
Record Dates: First submitted 2015-07-14; First posted 2015-08-17 (Estimated); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Graft vs Host Disease
Keywords: GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (20):
- Arm 1: Phase 1 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 1: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2A: Phase 1 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2A: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2A: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2B: Phase 1 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2B: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2 (Experimental): Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Interventions: Drug: Pregnyl®
- Arm 1: Phase 2 MTD (Experimental): After completion of the dose finding trial for each arm, the final doses will be carried forward into a two-stage phase II extension trial to confirm safety and make a preliminary determination of the activity level for Arm 1 and Arm 2. If the phase I trial enrolls fewer than 13 patients at the MTD, we will employ Simon's Minmax two-stage design with the possibility to discontinue after the 1st stage if the response rate is low
  Interventions: Drug: Pregnyl®
- Arm 2A: MTD (Experimental): After completion of the dose finding trial for each arm, the final doses will be carried forward into a two-stage phase II extension trial to confirm safety and make a preliminary determination of the activity level for Arm 1 and Arm 2. If the phase I trial enrolls fewer than 13 patients at the MTD, we will employ Simon's Minmax two-stage design with the possibility to discontinue after the 1st stage if the response rate is low
  Interventions: Drug: Pregnyl®
- Arm 2B: MTD (Experimental): After completion of the dose finding trial for each arm, the final doses will be carried forward into a two-stage phase II extension trial to confirm safety and make a preliminary determination of the activity level for Arm 1 and Arm 2. If the phase I trial enrolls fewer than 13 patients at the MTD, we will employ Simon's Minmax two-stage design with the possibility to discontinue after the 1st stage if the response rate is low
  Interventions: Drug: Pregnyl®

INTERVENTIONS:
Drug: Pregnyl® — Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
  Other Names: Human chorionic gonadotropin (hCG)

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of Pregnyl® when given in combination with standard immunosuppressive therapy in pediatric and adult patients with high-risk (Arm 1) or refractory/dependent (Arm 2) aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* Acute graft versus host disease (GVHD) fitting one of the following categories:

  * High-Risk aGVHD (ARM 1): Pediatric or adult (ages 12-76 years) HCT recipients with high-risk acute GVHD, as determined by the refined MN acute GVHD risk score: http://z.umn.edu/MNAcuteGVHDRiskScore OR high risk on the basis of blood biomarkers (Ann Arbor Score 3 or amphiregulin ≥ 33 pg/ml) or
  * Steroid-Refractory aGVHD (ARM 2): Pediatric or adult (ages 12-76 years) HCT recipient with grade II-IV steroid refractory or steroid-dependent acute GVHD, defined as any one of the following:

    * No response of acute GVHD after at least 4 days of systemic corticosteroids of at least 2 mg/kg prednisone or equivalent
    * Progression of acute GVHD within 3 days of systemic corticosteroids of at least 2 mg/kg prednisone or equivalent
    * Failure to improve to at least grade II acute GVHD after 14 days of systemic corticosteroids, with initial doses of at least 2 mg/kg prednisone or equivalent
    * Flare of acute GVHD of at least grade II/IV severity despite tapering dose of steroids being > 0.5 mg/kg/day.
* Adequate organ function at study enrollment defined as:

  * Renal: 1.73m2Serum creatinine ≤2.5x upper limit of normal (ULN)
  * Cardiac: Left ventricular ejection fraction (LVEF) ≥ 35%
* Voluntary written consent (adult or parent/guardian with minor assent for 12 through 17 year olds)

Exclusion Criteria:

* Progressive malignancy
* Diagnosis of a hormone responsive malignancy
* Uncontrolled infection at initiation of protocol treatment
* Current thromboembolic disease requiring full-dose anticoagulation - patients receiving pharmacologic prophylaxis for thromboembolic disease will be eligible
* Active or recent (within prior 3 months) thrombus, irrespective of anticoagulation status
* Pregnancy as assessed on baseline blood hCG level
* Unwilling or unable to stop supplemental sex hormone therapy (estrogen, progesterone, and/or testosterone preparations)
* Women or men of childbearing potential unwilling to take adequate precautions to avoid pregnancy from the start of protocol treatment through 28 days after the last treatment

Screening Inclusion Criteria:

* Pediatric or adult (ages 0-76 years) HCT recipients
* Suspected high risk GVHD
* Voluntary written consent (adult or parent/guardian with minor assent for 12 through 17 year olds)

Max Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shernan Holtan, MD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Holtan SG, Hoeschen A, Cao Q, Ustun C, Betts BC, Jurdi NE, Maakaron J, Rashidi A, Miller JS, Wagner JE, Blazar BR, Jacobson PA, Panoskaltsis-Mortari A, Weisdorf DJ, MacMillan ML. Phase II, Open-Label Clinical Trial of Urinary-Derived Human Chorionic Gonadotropin/Epidermal Growth Factor for Life-Threatening Acute Graft-versus-Host Disease. Transplant Cell Ther. 2023 Aug;29(8):509.e1-509.e8. doi: 10.1016/j.jtct.2023.05.021. Epub 2023 Jun 4. PMID 37279855
- [Derived] Holtan SG, Hoeschen AL, Cao Q, Arora M, Bachanova V, Brunstein CG, Miller JS, Rashidi A, Slungaard A, Ustun C, Vercellotti GM, Warlick ED, Betts BC, El Jurdi N, He F, Chen C, Gandhi I, Wagner JE, Blazar BR, Jacobson PA, Shabaneh A, Wang J, Panoskaltsis-Mortari A, MacMillan ML, Weisdorf DJ. Facilitating resolution of life-threatening acute GVHD with human chorionic gonadotropin and epidermal growth factor. Blood Adv. 2020 Apr 14;4(7):1284-1295. doi: 10.1182/bloodadvances.2019001259. PMID 32236525

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Phase 2 Dose Level -2: 125 USP hCG/875 pg EGF/m^2; Arm 1: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2; Arm 1: Phase 2 Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2; Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 1: Phase 2 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 1: Phase 2 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
- Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2A: Phase 1 Dose Level -2: 125 USP hCG/875 pg EGF/m^2; Arm 2A: Phase 2 Dose Level -2: 125 USP hCG/875 pg EGF/m^2; Arm 2A: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2; Arm 2A: Phase 2 Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2; Arm 2A: Phase 2 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 2A: Phase 2 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
- Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2B: Phase 1 Dose Level -2: 125 USP hCG/875 pg EGF/m^2; Arm 2B: Phase 2 Dose Level -2: 125 USP hCG/875 pg EGF/m^2; Arm 2B: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2; Arm 2B: Phase 2 Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 2B: Phase 2 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2B: Phase 2 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2B: Phase 2 Dose Level 3 2,000 USP; Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2; Arm 2B: Phase 2 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2; Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m; Arm 2B: Phase 2 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
Period: Overall Study
Arm/Group | Arm 1: Phase 1 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 | Arm 1: Phase 2 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 | Arm 1: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 | Arm 1: Phase 2 Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2A: Phase 1 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 | Arm 2A: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2B: Phase 1 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level -2: 125 USP hCG/875 pg EGF/m^2 | Arm 2B: Phase I Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level -1: 250 USP hCG/1,750 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2 | Arm 2B: Phase 2 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m | Arm 2B: Phase 2 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m
Started | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 9 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 8 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 5 | 1 | 2 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 9 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 8 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5 | 1 | 2 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2; Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2; Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has toxicity that meets the definition of dose limiting, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m | Total
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3 | 53
Age, Continuous [Median (Full Range); unit: Years] | 46 [39 to 53] | 64 [64 to 64] | 60.5 [22 to 72] | 60.5 [22 to 72] | 57 [57 to 57] | 61.5 [26 to 67] | 61.5 [26 to 67] | 56.5 [50 to 63] | 63 [63 to 63] | 64 [35 to 66] | 64 [35 to 66] | 61 [53 to 69] | 50 [2 to 55] | 61 [2 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 3 | 0 | 1 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 14
  Male | 2 | 1 | 6 | 10 | 1 | 3 | 5 | 1 | 1 | 4 | 0 | 2 | 3 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 1 | 2 | 9 | 13 | 1 | 4 | 7 | 2 | 1 | 5 | 1 | 2 | 2 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 1 | 1 | 8 | 12 | 1 | 3 | 7 | 2 | 1 | 5 | 0 | 2 | 3 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3 | 53

OUTCOME MEASURES:

1. Primary Outcome: Phase I: MTD (USP hCG)
Description: Maximum tolerated dose (MTD) of Pregnyl® when given with standard immunosuppressive therapy in pediatric and adult patients with high-risk or refractory acute graft-versus-host disease (aGVHD). Dosage measured as (USP hCG/pg EGF/mm^2).
Time Frame: Day 14 after initiation of protocol therapy
Measure: Number; unit: Pregnyl dosage (USP hCG)
Groups:
- 1: High-Risk aGVHD: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has toxicity that meets the definition of dose limiting, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m2
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
- 2a: Steroid-Dependent aGVHD: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m2
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
- 2b: Steroid-Refractory aGVHD: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m2
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
Arm/Group | 1: High-Risk aGVHD | 2a: Steroid-Dependent aGVHD | 2b: Steroid-Refractory aGVHD
Number analyzed (Participants) | 26 | 13 | 12
Pregnyl dosage (USP hCG) | 2000 | 2000 | 5000

2. Primary Outcome: Phase I: MTD (pg EGF/m^2)
Description: Maximum tolerated dose (MTD) of Pregnyl® when given with standard immunosuppressive therapy in pediatric and adult patients with high-risk or refractory acute graft-versus-host disease (aGVHD). Dosage measured as (USP hCG/pg EGF/m^2).
Time Frame: Day 14 after initiation of protocol therapy
Measure: Number; unit: Pregnyl dosage (pg EGF/m^2)
Arm/Group | 1: High-Risk aGVHD | 2a: Steroid-Dependent aGVHD | 2b: Steroid-Refractory aGVHD
Number analyzed (Participants) | 26 | 13 | 12
Pregnyl dosage (pg EGF/m^2) | 14000 | 14000 | 34000

3. Primary Outcome: Number of Patients With Complete Response
Description: Percentage of complete response among surviving patients at day 28 after initiation of protocol therapy in pediatric and adult patients with high-risk (Arm 1) or refractory (Arm 2) aGVHD. Complete response is defined as a Stage of 0 for all organs with no additional intervening therapy for their GVHD.
Time Frame: Day 28 after initiation of protocol therapy
Measure: Number; unit: participants
Groups:
- Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
- Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
participants | 2 | 2 | 4 | 7 | 1 | 3 | 5 | 1 | 0 | 2 | 0 | 0 | 1

4. Primary Outcome: Number of Patients With Partial Response
Description: Percentage of partial response among surviving patients at day 28 after initiation of protocol therapy in pediatric and adult patients with high-risk (Arm 1) or refractory (Arm 2) aGVHD. Partial response is defined as improvement by at least 1 stage in all involved organs without progression in others with no additional intervening therapy for their GVHD.
Time Frame: Day 28 after initiation of protocol therapy
Measure: Number; unit: participants
Groups:
- Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
participants | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1

5. Primary Outcome: Number of Patients With Mixed Response
Description: Percentage of mixed response among surviving patients at day 28 after initiation of protocol therapy in pediatric and adult patients with high-risk (Arm 1) or refractory (Arm 2) aGVHD. Mixed Response is defined as improvement in one organ with deterioration in another organ manifesting symptoms of GVHD or development of symptoms of GVHD in a new organ.
Time Frame: Day 28 after initiation of protocol therapy
Measure: Number; unit: participants
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
participants | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0

6. Primary Outcome: Number of Patients With No Response
Description: Percentage of no response among surviving patients at day 28 after initiation of protocol therapy in pediatric and adult patients with high-risk (Arm 1) or refractory (Arm 2) aGVHD. No response is defined as deterioration of any organ involved.
Time Frame: Day 28 after initiation of protocol therapy
Measure: Number; unit: participants
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
participants | 0 | 0 | 4 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1

7. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Feasibility of hCG Supplementation With Pregnyl®
Description: Safety and feasibility of hCG supplementation with Pregnyl® in combination with standard immunosuppressive therapy in pediatric and adult patients with high-risk or refractory aGVHD.
Time Frame: Day 70 after initiation of protocol therapy
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
- Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
- Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2; Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has toxicity that meets the definition of dose limiting, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
Participants | 1 | 1 | 3 | 6 | 1 | 2 | 5 | 2 | 1 | 3 | 1 | 2 | 1

8. Secondary Outcome: Number of Participants With Incidence of aGVHD Flare
Description: Incidence of acute GVHD flare after CR/PR requiring increase of steroids or other systemic treatment at day 28.
Time Frame: Day 28 after initiation of protocol therapy
Measure: Number; unit: participants
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
participants | 0 | 0 | 3 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1

9. Secondary Outcome: Number of Participants With Incidence of aGVHD Flare
Description: Incidence of acute GVHD flare after CR/PR requiring increase of steroids or other systemic treatment at day 56.
Time Frame: Day 56 after initiation of protocol therapy
Measure: Number; unit: participants
Groups:
- Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2; Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
participants | 0 | 0 | 2 | 8 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 1

10. Secondary Outcome: Rate of Participants Who Fail Treatment at Day 28
Description: Rate of treatment failure for acute GVHD at day 28 after initiation of protocol therapy to historical controls.
Time Frame: Day 28 after initiation of protocol therapy
Measure: Number; unit: participants
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
participants | 0 | 0 | 8 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 1

11. Secondary Outcome: Rate of Participants Who Fail Treatment at Day 56
Description: Rate of treatment failure for acute GVHD at day 56 after initiation of protocol therapy to historical controls.
Time Frame: Day 56 after initiation of protocol therapy
Measure: Number; unit: participants
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m^2
Number analyzed (Participants) | 2 | 2 | 9 | 13 | 1 | 4 | 8 | 2 | 1 | 5 | 1 | 2 | 3
participants | 0 | 0 | 2 | 9 | 0 | 2 | 4 | 1 | 0 | 2 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: 70 Days after first treatment
Groups:
- Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 7 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort has reached day 21 to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has a toxicity, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
- Arm 2B: Phase 2 Dose Level 3 2,000 USP; Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2; Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m: Standard of care immunosuppression, plus Pregnyl® (hCG supplementation) at assigned dose subcutaneously every other day for up to 5 doses of Pregnyl®; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic.
  The 1st 2 patients will be enrolled in dose level 1. The next cohort of 2 patients will not begin treatment until all patients in the current cohort have reached day 21 in order to assess for dose limiting toxicity (DLT).
  Individual patient dose reductions: If a patient has toxicity that meets the definition of dose limiting, the patient can drop down one dose level for the next injection and continue treatment.
  Pregnyl®: Standard of care immunosuppression, plus Pregnyl® at assigned dose subcutaneously every other day for up to 5 doses through day 7
  Phase I: up to 7 dose levels of Pregnyl® will be tested; however dose levels -1 and -2 will be used only if dose level 1 proves too toxic. Study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD).
  Step -2: 125 USP hCG/875 pg EGF/m2 Step -1: 250 USP hCG/1,750 pg EGF/m2 Step 1 (start): 500 USP hCG/3,500 pg EGF/m2 Step 2: 1,000 USP hCG/7,000 pg EGF/m2 Step 3: 2,000 USP hCG/14,000 pg EGF/m2 Step 4 (Arm 2b only): 3,500 USP hCG/24,500 pg EGF/m2 Step 5 (Arm 2b only): 5,000 USP hCG/35,000 pg EGF/m
  Phase II: the dose of Pregnyl will be that identified as the MTD during phase I.
Arm/Group | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 | Arm 2B: Phase 2 Dose Level 3 2,000 USP | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2 | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/2 | 0/9 | 0/13 | 0/1 | 1/4 | 0/8 | 0/2 | 1/1 | 0/5 | 1/1 | 1/2 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 1/9 | 2/13 | 1/1 | 2/4 | 4/8 | 2/2 | 1/1 | 5/5 | 0/1 | 2/2 | 3/3
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 3/9 | 6/13 | 1/1 | 2/4 | 5/8 | 2/2 | 1/1 | 3/5 | 1/1 | 2/2 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 (N=2) | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (N=2) | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=9) | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=13) | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (N=1) | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=4) | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=8) | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 (N=2) | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (N=1) | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=5) | Arm 2B: Phase 2 Dose Level 3 2,000 USP (N=1) | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2 (N=2) | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m (N=3)
blood and lympathic system (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duode0l obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duode0l perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointesti0l disorders - Other, (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible posterior (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 (N=2) | Arm 1: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (N=2) | Arm 1: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=9) | Arm 1: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=13) | Arm 2A: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (N=1) | Arm 2A: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=4) | Arm 2A: Phase 2 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=8) | Arm 2B: Phase 1 Dose Level 1 500 USP hCG/3,500 pg EGF/m^2 (N=2) | Arm 2B: Phase 1 Dose Level 2 1,000 USP hCG/7,000 pg EGF/m^2 (N=1) | Arm 2B: Phase 1 Dose Level 3 2,000 USP hCG/14,000 pg EGF/m2 (N=5) | Arm 2B: Phase 2 Dose Level 3 2,000 USP (N=1) | Arm 2B: Phase 1 Dose Level 4 3,500 USP hCG/24,500 pg EGF/m2 (N=2) | Arm 2B: Phase 1 Dose Level 5 5,000 USP hCG/35,000 pg EGF/m (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (10) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT02525029/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT02525029/ICF_001.pdf